CLINICAL TRIAL: NCT02864654
Title: Effectiveness and Safety of Adipose-Derived Regenerative Cells for the Treatment of Critical Lower Limb Ischemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Central Clinical Hospital w/Outpatient Health Center of Business Administration for the President of Russian Federation (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RU-CCH-07-01-16
Record Dates: First submitted 2016-08-05; First posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Critical Limb Ischemia; Arteriosclerosis Obliterans; Peripheral Arterial Disease; Thromboangiitis Obliterans; Diabetic Angiopathies
Keywords: Critical lower limb ischemia; Atherosclerosis obliterans; Diabetic angiopathies; Thromboangiitis obliterans; Ischemic ulcers; Peripheral arterial disease; Indirect revascularisation; Intramuscular injection; Ankle-brachial index; Transcutaneous oxygen tension; Stromal vascular fraction (SVF); Adipose-derived regenerative cells (ADRC); Adipose tissue; Stem cells
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Arteriosclerosis Obliterans; Peripheral Arterial Disease; Thromboangiitis Obliterans; Diabetic Angiopathies | interventions — Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADRC injection (Experimental): Subjects will undergo liposuction under local anesthesia. Lipoaspirate will be processed to isolate and concentrate Adipose-derived regenerative cells (ADRC). After isolation 10 mL of autologous ADRC suspension will be injected intramuscularly, close to the site of muscle injury. 10 to 20 injections will be performed so as to infiltrate the injured muscle
  Interventions: Procedure: ADRC injection; Other: ADRC isolation; Procedure: Liposuction

INTERVENTIONS:
Procedure: ADRC injection — 10 mL of autologous ADRC suspension will be injected intramuscularly
Other: ADRC isolation — ADRC will be isolated according to patent pending technology based on enzymatic digestion, washing and concentration of cell pellet in 10 ml of normal saline.
Procedure: Liposuction

SUMMARY:
Adipose-derived regenerative cells (ADRC) will be extracted from lipoaspirate by enzymatic digestion. 10 mL of autologous ADRC suspension injected intramuscularly, close to the site of muscle injury. All patients will receive cell therapy. This is a single arm study with no control.

DETAILED DESCRIPTION:
Fat tissue obtainment:

Subjects will undergo liposuction under local anesthesia. In this procedure, Ringer's solution with the anesthetic lidocaine and vasoconstrictor adrenaline infused into the adipose compartment to minimize blood loss and contamination of the tissue by peripheral blood cells. 15 minutes later a hollow blunt-tipped 3 mm cannula introduced into the subcutaneous space through small (0.5 cm) incision. The cannula attached to syringe and under gentle suction moved through the adipose compartment, mechanically disrupting the fat tissue. Aspirate volume - approximately 150-200 cc. Procedure time - 30 minutes.

ADRC isolation:

Harvested adipose tissue will be processed according to patent pending technology based on enzymatic digestion, washing and concentration of cell pellet in 10.5 ml of normal saline. Obtained ADRC divided into 2 portions. First portion (0.5 mL) used for counting, viability and sterility assessment. The second portion (10 ml) placed into sterile syringe for injection.

Autologous ADRC administration

10 mL of autologous ADRC suspension will be injected intramuscularly, close to the site of muscle injury. 10 to 20 injections (0.5 to 1.0 mL each) will be performed so as to infiltrate the injured muscle.

ELIGIBILITY:
Inclusion Criteria:

* Patients with critical lower limb ischemia, with resting pain wich can't be adequately managed by opioid analgetics and/or foot ulcers or necrosis, with II-4, III-5 и IV-6 stages of chronic arterial failure according to Rutherford's classification
* Ankle-brachial index less than 0.4 and/or ТСрО2 less than 30 mm Hg
* Patients with lower limbs' arteries lesions revealed by angiography uneffectiveness or impossibility of limb's revascularisation or patient's refusal of the procedure
* Patient is familiar with Participant information sheet
* Patient signed informed consent form

Non-inclusion Criteria:

* Contraindications for local anesthesia or history of allergy for local anesthetics
* Systemic glucocorticoid and/or immunosuppressant therapy
* Any condition that might limit compliance (dementia, mental disorders, narcotic drug or alcohol abuse etc.)
* Participation in other clinical trials (or administration of investigational drugs) during 3 months prior inclusion
* Patients with malignant tumors including postoperative period, patients receiving chemotherapy and/or radiotherapy
* Clinically significant abnormalities in results of laboratory tests
* Patient received anticoagulants at least 12 hours prior the liposuction
* Medical history of heterotopic ossifications
* Patients prescribed for glycoprotein inhibitors treatment

Exclusion Criteria:

* Patient's refusal from the further participation in trial
* Chronic kidney disease IV- V stages (creatinine clearance < 30 mL/min estimated by Cockcroft-Gault formula)
* Confirmed syphilis, HIV, hepatitis B or C infections

Dropout Criteria:

* Indications for the amputation of the limb

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-08 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Serious adverse events | 4 weeks after injection of ADRC suspension
  Frequency, type and severity of serious adverse events (SAE)
Serious adverse reactions | 4 weeks after injection of ADRC suspension
  Frequency, type and severity of serious adverse reactions (SAR)

SECONDARY OUTCOMES:
Changes of ankle-brachial index | Follow up to completion (24 weeks after intervention)
  Influence of intervention on ankle-brachial index.
Changes of hemodynamics in lower extremity - 1 | Follow up to completion (24 weeks after intervention)
  Influence of intervention on blood flow velocity assessed by arterial duplex scanning.
Changes of hemodynamics in lower extremity - 2 | Follow up to completion (24 weeks after intervention)
  Influence of intervention on pulsatility index assessed by arterial duplex scanning.
Changes of hemodynamics in lower extremity - 3 | Follow up to completion (24 weeks after intervention)
  Influence of intervention on resistance index assessed by arterial duplex scanning.
Metabolic state of targeted tissues measurements | Follow up to completion (24 weeks after intervention)
  Changes of transcutaneous oxygen tension (ТсРО2) in injured limb assessed by transcutaneous oximetry.
Quality of life monitoring - 1 | Follow up to completion (24 weeks after intervention)
  Quality of life estimated by validated questionnaire: the Short Form (SF-36).
Quality of life monitoring - 2 | Follow up to completion (24 weeks after intervention)
  Quality of life estimated by validated questionnaire:Peripheral Artery Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Andrey A Kalinin, MD, PhD, Principal Investigator — Federal State Budgetary Institution "Central Clinical Hospital with Outpatient Health Center" of the Business Administration for the President of the Russian Federation; Andrey A Pulin, MD, PhD, Principal Investigator — Federal State Budgetary Institution "Central Clinical Hospital with Outpatient Health Center" of the Business Administration for the President of the Russian Federation; Evgeny R Lysenko, MD, PhD, Prof, Study Director — FSBI Federal Clinial Center of Advanced medical Technologies FMBA of Russia
Locations (1):
- Federal State Budgetary Institution "Central Clinical Hospital with Outpatient Health Center" of the Business Administration for the President of the Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided